CLINICAL TRIAL: NCT00074373
Title: The Research Registry for Neonatal Lupus
Status: Completed | Type: Observational
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Other Study IDs: 09-0289
Record Dates: First submitted 2003-12-11; First posted 2003-12-12 (Estimated); Last update posted 2023-08-03 (Actual); Status verified 2023-08

CONDITIONS: Neonatal Lupus; Systemic Lupus Erythematosus; Sjogren's Syndrome; Congenital Heart Block
Keywords: Anti-SSA/Ro Antibodies; Anti-SSB/La Antibodies
MeSH Terms: conditions — Neonatal Systemic lupus erythematosus; Lupus Erythematosus, Systemic; Sjogren's Syndrome; Congenital heart block

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- human beings: human beings of all sexes, ages, and health statuses
  Interventions: Other: No intervention; observational

INTERVENTIONS:
Other: No intervention; observational
  Other Names: The study is observational

SUMMARY:
Women with lupus and other related disorders produce certain antibodies in the blood. Some women have these antibodies even if they have not yet developed symptoms of lupus or Sjogren's syndrome. When these women become pregnant, they may pass the antibodies to their infants. The infants may then develop a disease called neonatal lupus. The symptoms of neonatal lupus include an abnormally slow heart beat (heart block) and a skin rash. This registry collects information on women and infants affected by neonatal lupus as well as other family members who may be healthy.

DETAILED DESCRIPTION:
Neonatal lupus is a disease seen in babies born to mothers who have antibodies to SSA/Ro and/or SSB/La proteins. The mother may have systemic lupus erythematosus, Sjogren's syndrome, or be otherwise healthy. Heart block and a characteristic skin rash are the primary manifestations of neonatal lupus.

The Research Registry for Neonatal Lupus was initiated in 1994 to help basic scientists and clinicians better understand the cause of neonatal lupus and discover a cure. The Research Registry is a central repository of patient information, sera, and DNA. The Registry provides blood samples (kept anonymous) to scientists studying neonatal lupus. Information from the registry forms the basis of family counseling and tracks important data such as recurrence rates in subsequent pregnancies and the effects of treatments. The Research Registry also serves as an educational resource for women who are eager to learn about this disease.

Women with a child affected by neonatal lupus may enroll in the Registry. Women can be self referred or referred by their doctors. Siblings of women with a child affected by neonatal lupus, fathers and maternal grandparents of children with neonatal lupus, and unaffected siblings of a child with neonatal lupus are also invited to participate in this study. All information on the mother and her family is confidential; only nonidentifying information will be provided to researchers. Women interested in the registry will be sent articles and educational materials about neonatal lupus, a consent form for the Registry, and an enrollment questionnaire. Participants will be asked to sign a medical records release form. Participants will also be asked to donate a blood sample for antibody testing and DNA isolation.

ELIGIBILITY:
Inclusion Criteria:

* Mother with antibodies to SSA/Ro, SSB/La, or ribonucleoproteins (RNP) OR Child of mother with such antibodies who has neonatal lupus (congenital heart block, transient skin rash, and/or hepatic or hematologic manifestations) OR Father of neonatal lupus-affected child OR Maternal grandparents of neonatal lupus-affected child OR Maternal aunts and uncles of neonatal lupus-affected OR Unaffected siblings of neonatal lupus-affected child

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Women with a child affected by neonatal lupus, children affected by neonatal lupus, siblings of children affected by neonatal lupus, siblings of women with a child affected by neonatal lupus, fathers and maternal grandparents of children with neonatal lupus, and unaffected people to serve as controls are invited to participate in this study.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2010-05-27 (Actual); Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
means of curing and/or preventing neonatal lupus | ongoing
  means of curing and/or preventing neonatal lupus

SECONDARY OUTCOMES:
identification of pathogenesis of neonatal lupus | ongoing
  identification of pathogenesis of neonatal lupus

CONTACTS AND LOCATIONS:
Overall Officials: Jill P. Buyon, MD, Study Director — NYU Medical Center, NYU School of Medicine
Locations (1):
- Jill P. Buyon, MD, New York, New York, United States

REFERENCES:
- [Background] Buyon JP, Clancy RM. Neonatal lupus: review of proposed pathogenesis and clinical data from the US-based Research Registry for Neonatal Lupus. Autoimmunity. 2003 Feb;36(1):41-50. doi: 10.1080/0891693031000067340. PMID 12765470
- [Background] Solomon DG, Rupel A, Buyon JP. Birth order, gender and recurrence rate in autoantibody-associated congenital heart block: implications for pathogenesis and family counseling. Lupus. 2003;12(8):646-7. doi: 10.1191/0961203303lu425xx. No abstract available. PMID 12945727
- [Background] Askanase AD, Miranda-Carus ME, Tang X, Katholi M, Buyon JP. The presence of IgG antibodies reactive with components of the SSA/Ro-SSB/La complex in human breast milk: implications in neonatal lupus. Arthritis Rheum. 2002 Jan;46(1):269-71. doi: 10.1002/1529-0131(200201)46:13.0.CO;2-6. No abstract available. PMID 11817601
- [Background] Askanase AD, Friedman DM, Copel J, Dische MR, Dubin A, Starc TJ, Katholi MC, Buyon JP. Spectrum and progression of conduction abnormalities in infants born to mothers with anti-SSA/Ro-SSB/La antibodies. Lupus. 2002;11(3):145-51. doi: 10.1191/0961203302lu173oa. PMID 11999879
- [Background] Martin V, Lee LA, Askanase AD, Katholi M, Buyon JP. Long-term followup of children with neonatal lupus and their unaffected siblings. Arthritis Rheum. 2002 Sep;46(9):2377-83. doi: 10.1002/art.10638. PMID 12355485
- [Background] Neiman AR, Lee LA, Weston WL, Buyon JP. Cutaneous manifestations of neonatal lupus without heart block: characteristics of mothers and children enrolled in a national registry. J Pediatr. 2000 Nov;137(5):674-80. doi: 10.1067/mpd.2000.109108. PMID 11060534
- [Background] Buyon JP, Hiebert R, Copel J, Craft J, Friedman D, Katholi M, Lee LA, Provost TT, Reichlin M, Rider L, Rupel A, Saleeb S, Weston WL, Skovron ML. Autoimmune-associated congenital heart block: demographics, mortality, morbidity and recurrence rates obtained from a national neonatal lupus registry. J Am Coll Cardiol. 1998 Jun;31(7):1658-66. doi: 10.1016/s0735-1097(98)00161-2. PMID 9626848
- [Background] Clancy RM, Buyon JP. Autoimmune-associated congenital heart block: dissecting the cascade from immunologic insult to relentless fibrosis. Anat Rec A Discov Mol Cell Evol Biol. 2004 Oct;280(2):1027-35. doi: 10.1002/ar.a.20072. PMID 15368347
- [Background] Clancy RM, Buyon JP. More to death than dying: apoptosis in the pathogenesis of SSA/Ro-SSB/La-associated congenital heart block. Rheum Dis Clin North Am. 2004 Aug;30(3):589-602, x. doi: 10.1016/j.rdc.2004.04.013. PMID 15261343
- [Background] Clancy RM, Kapur RP, Molad Y, Askanase AD, Buyon JP. Immunohistologic evidence supports apoptosis, IgG deposition, and novel macrophage/fibroblast crosstalk in the pathologic cascade leading to congenital heart block. Arthritis Rheum. 2004 Jan;50(1):173-82. doi: 10.1002/art.11430. PMID 14730614
- [Background] Hu K, Qu Y, Yue Y, Boutjdir M. Functional basis of sinus bradycardia in congenital heart block. Circ Res. 2004 Mar 5;94(4):e32-8. doi: 10.1161/01.RES.0000121566.01778.06. Epub 2004 Feb 12. PMID 14963005
- [Background] Clancy RM, Backer CB, Yin X, Chang MW, Cohen SR, Lee LA, Buyon JP. Genetic association of cutaneous neonatal lupus with HLA class II and tumor necrosis factor alpha: implications for pathogenesis. Arthritis Rheum. 2004 Aug;50(8):2598-603. doi: 10.1002/art.20442. PMID 15334474
- [Background] Gordon P, Khamashta MA, Rosenthal E, Simpson JM, Sharland G, Brucato A, Franceschini F, De Bosschere K, Meheus L, Meroni PL, Hughes GR, Buyon J. Anti-52 kDa Ro, anti-60 kDa Ro, and anti-La antibody profiles in neonatal lupus. J Rheumatol. 2004 Dec;31(12):2480-7. PMID 15570655
- [Background] Glickstein J, Buyon J, Kim M, Friedman D; PRIDE investigators. The fetal Doppler mechanical PR interval: a validation study. Fetal Diagn Ther. 2004 Jan-Feb;19(1):31-4. doi: 10.1159/000074256. PMID 14646414
- [Background] Tran HB, Cavill D, Buyon JP, Gordon TP. Intravenous immunoglobulin and placental transport of anti-Ro/La antibodies: comment on the letter by Kaaja and Julkunen. Arthritis Rheum. 2004 Jan;50(1):337-8; author reply 338. doi: 10.1002/art.11498. No abstract available. PMID 14730639
- [Background] Buyon JP, Rupel A, Clancy RM. Neonatal lupus syndromes. Lupus. 2004;13(9):705-12. doi: 10.1191/0961203304lu2008oa. PMID 15485109
- [Background] Neufing PJ, Clancy RM, Jackson MW, Tran HB, Buyon JP, Gordon TP. Exposure and binding of selected immunodominant La/SSB epitopes on human apoptotic cells. Arthritis Rheum. 2005 Dec;52(12):3934-42. doi: 10.1002/art.21486. PMID 16320341
- [Background] Clancy RM, Buyon JP, Ikeda K, Nozawa K, Argyle DA, Friedman DM, Chan EK. Maternal antibody responses to the 52-kd SSA/RO p200 peptide and the development of fetal conduction defects. Arthritis Rheum. 2005 Oct;52(10):3079-86. doi: 10.1002/art.21289. PMID 16200587
- [Background] Buyon JP, Clancy RM. Autoantibody-associated congenital heart block: TGFbeta and the road to scar. Autoimmun Rev. 2005 Jan;4(1):1-7. doi: 10.1016/j.autrev.2004.04.003. PMID 15652772
- [Background] Kamel R, Eftekhari P, Clancy R, Buyon JP, Hoebeke J. Autoantibodies against the serotoninergic 5-HT4 receptor and congenital heart block: a reassessment. J Autoimmun. 2005 Aug;25(1):72-6. doi: 10.1016/j.jaut.2005.04.005. PMID 16009533
- [Background] Buyon JP, Askanase AD, Kim MY, Copel JA, Friedman DM. Identifying an early marker for congenital heart block: when is a long PR interval too long? Comment on the article by Sonesson et al. Arthritis Rheum. 2005 Apr;52(4):1341-2. doi: 10.1002/art.20971. No abstract available. PMID 15818705
- [Background] Buyon JP, Clancy RM. Neonatal lupus: basic research and clinical perspectives. Rheum Dis Clin North Am. 2005 May;31(2):299-313, vii. doi: 10.1016/j.rdc.2005.01.010. PMID 15922147
- [Background] Stea EA, Routsias JG, Clancy RM, Buyon JP, Moutsopoulos HM, Tzioufas AG. Anti-La/SSB antiidiotypic antibodies in maternal serum: a marker of low risk for neonatal lupus in an offspring. Arthritis Rheum. 2006 Jul;54(7):2228-34. doi: 10.1002/art.21954. PMID 16802359
- [Background] Askanase AD, Iloh I, Buyon JP. Hypothyroidism and antithyroglobulin and antithyroperoxidase antibodies in the pathogenesis of autoimmune associated congenital heart block. J Rheumatol. 2006 Oct;33(10):2099. No abstract available. PMID 17014028
- [Background] Bachmann MP, Bartsch H, Gross JK, Maier SM, Gross TF, Workman JL, James JA, Farris AD, Jung B, Franke C, Conrad K, Schmitz M, Buttner C, Buyon JP, Semsei I, Harley JB, Rieber EP. Autoimmunity as a result of escape from RNA surveillance. J Immunol. 2006 Aug 1;177(3):1698-707. doi: 10.4049/jimmunol.177.3.1698. PMID 16849479
- [Background] Clancy RM, Neufing PJ, Zheng P, O'Mahony M, Nimmerjahn F, Gordon TP, Buyon JP. Impaired clearance of apoptotic cardiocytes is linked to anti-SSA/Ro and -SSB/La antibodies in the pathogenesis of congenital heart block. J Clin Invest. 2006 Sep;116(9):2413-22. doi: 10.1172/JCI27803. Epub 2006 Aug 10. PMID 16906225
- [Background] Clancy RM, Zheng P, O'Mahony M, Izmirly P, Zavadil J, Gardner L, Buyon JP. Role of hypoxia and cAMP in the transdifferentiation of human fetal cardiac fibroblasts: implications for progression to scarring in autoimmune-associated congenital heart block. Arthritis Rheum. 2007 Dec;56(12):4120-31. doi: 10.1002/art.23061. PMID 18050204
- [Background] Izmirly PM, Rivera TL, Buyon JP. Neonatal lupus syndromes. Rheum Dis Clin North Am. 2007 May;33(2):267-85, vi. doi: 10.1016/j.rdc.2007.02.005. PMID 17499707
- [Background] Friedman DM, Rupel A, Buyon JP. Epidemiology, etiology, detection, and treatment of autoantibody-associated congenital heart block in neonatal lupus. Curr Rheumatol Rep. 2007 May;9(2):101-8. doi: 10.1007/s11926-007-0003-4. PMID 17502039
- [Background] Rivera TL, Izmirly PM, Birnbaum BK, Byrne P, Brauth JB, Katholi M, Kim MY, Fischer J, Clancy RM, Buyon JP. Disease progression in mothers of children enrolled in the Research Registry for Neonatal Lupus. Ann Rheum Dis. 2009 Jun;68(6):828-35. doi: 10.1136/ard.2008.088054. Epub 2008 Jul 14. PMID 18625627
- [Background] Strandberg L, Winqvist O, Sonesson SE, Mohseni S, Salomonsson S, Bremme K, Buyon JP, Julkunen H, Wahren-Herlenius M. Antibodies to amino acid 200-239 (p200) of Ro52 as serological markers for the risk of developing congenital heart block. Clin Exp Immunol. 2008 Oct;154(1):30-7. doi: 10.1111/j.1365-2249.2008.03732.x. Epub 2008 Aug 22. PMID 18727629
- [Background] Buyon JP, Brucato A, Friedman DM. What's in a name? Ann Rheum Dis. 2008 May;67(5):732; discussion 732. doi: 10.1136/ard.2007.082693. No abstract available. PMID 18408119
- [Background] Buyon JP, Clancy RM. Dying right to live longer: positing apoptosis as a link between maternal autoantibodies and congenital heart block. Lupus. 2008 Feb;17(2):86-90. doi: 10.1177/0961203307085115. PMID 18250129
- [Background] Niewold TB, Rivera TL, Buyon JP, Crow MK. Serum type I interferon activity is dependent on maternal diagnosis in anti-SSA/Ro-positive mothers of children with neonatal lupus. Arthritis Rheum. 2008 Feb;58(2):541-6. doi: 10.1002/art.23191. PMID 18240214
- [Background] Friedman DM, Kim MY, Copel JA, Davis C, Phoon CK, Glickstein JS, Buyon JP; PRIDE Investigators. Utility of cardiac monitoring in fetuses at risk for congenital heart block: the PR Interval and Dexamethasone Evaluation (PRIDE) prospective study. Circulation. 2008 Jan 29;117(4):485-93. doi: 10.1161/CIRCULATIONAHA.107.707661. Epub 2008 Jan 14. PMID 18195175
- [Background] Llanos C, Izmirly PM, Katholi M, Clancy RM, Friedman DM, Kim MY, Buyon JP. Recurrence rates of cardiac manifestations associated with neonatal lupus and maternal/fetal risk factors. Arthritis Rheum. 2009 Oct;60(10):3091-7. doi: 10.1002/art.24768. PMID 19790064
- [Background] Buyon JP, Clancy RM, Friedman DM. Autoimmune associated congenital heart block: integration of clinical and research clues in the management of the maternal / foetal dyad at risk. J Intern Med. 2009 Jun;265(6):653-62. doi: 10.1111/j.1365-2796.2009.02100.x. PMID 19493059
- [Background] Buyon JP, Clancy RM, Friedman DM. Cardiac manifestations of neonatal lupus erythematosus: guidelines to management, integrating clues from the bench and bedside. Nat Clin Pract Rheumatol. 2009 Mar;5(3):139-48. doi: 10.1038/ncprheum1018. PMID 19252519
- [Background] Friedman DM, Kim MY, Copel JA, Llanos C, Davis C, Buyon JP. Prospective evaluation of fetuses with autoimmune-associated congenital heart block followed in the PR Interval and Dexamethasone Evaluation (PRIDE) Study. Am J Cardiol. 2009 Apr 15;103(8):1102-6. doi: 10.1016/j.amjcard.2008.12.027. Epub 2009 Mar 4. PMID 19361597
- [Background] Llanos C, Chan EK, Li S, Abadal GX, Izmirly P, Byrne C, Clancy RM, Buyon JP. Antibody reactivity to alpha-enolase in mothers of children with congenital heart block. J Rheumatol. 2009 Mar;36(3):565-9. doi: 10.3899/jrheum.080860. Epub 2009 Feb 4. PMID 19208599
- [Background] Buyon JP. Updates on lupus and pregnancy. Bull NYU Hosp Jt Dis. 2009;67(3):271-5. PMID 19852749
- [Background] Briassouli P, Komissarova EV, Clancy RM, Buyon JP. Role of the urokinase plasminogen activator receptor in mediating impaired efferocytosis of anti-SSA/Ro-bound apoptotic cardiocytes: Implications in the pathogenesis of congenital heart block. Circ Res. 2010 Aug 6;107(3):374-87. doi: 10.1161/CIRCRESAHA.109.213629. Epub 2010 Jun 17. PMID 20558828
- [Background] Clancy RM, Alvarez D, Komissarova E, Barrat FJ, Swartz J, Buyon JP. Ro60-associated single-stranded RNA links inflammation with fetal cardiac fibrosis via ligation of TLRs: a novel pathway to autoimmune-associated heart block. J Immunol. 2010 Feb 15;184(4):2148-55. doi: 10.4049/jimmunol.0902248. Epub 2010 Jan 20. PMID 20089705
- [Background] Clancy RM, Marion MC, Kaufman KM, Ramos PS, Adler A; International Consortium on Systemic Lupus Erythematosus Genetics; Harley JB, Langefeld CD, Buyon JP. Identification of candidate loci at 6p21 and 21q22 in a genome-wide association study of cardiac manifestations of neonatal lupus. Arthritis Rheum. 2010 Nov;62(11):3415-24. doi: 10.1002/art.27658. PMID 20662065
- [Background] Askanase AD, Izmirly PM, Katholi M, Mumtaz J, Buyon JP. Frequency of neuro-psychiatric dysfunction in anti-SSA/SSB exposed children with and without neonatal lupus. Lupus. 2010 Mar;19(3):300-6. doi: 10.1177/0961203309354542. Epub 2009 Dec 14. PMID 20008445
- [Background] Friedman DM, Llanos C, Izmirly PM, Brock B, Byron J, Copel J, Cummiskey K, Dooley MA, Foley J, Graves C, Hendershott C, Kates R, Komissarova EV, Miller M, Pare E, Phoon CK, Prosen T, Reisner D, Ruderman E, Samuels P, Yu JK, Kim MY, Buyon JP. Evaluation of fetuses in a study of intravenous immunoglobulin as preventive therapy for congenital heart block: Results of a multicenter, prospective, open-label clinical trial. Arthritis Rheum. 2010 Apr;62(4):1138-46. doi: 10.1002/art.27308. PMID 20391423
- [Background] Izmirly PM, Llanos C, Lee LA, Askanase A, Kim MY, Buyon JP. Cutaneous manifestations of neonatal lupus and risk of subsequent congenital heart block. Arthritis Rheum. 2010 Apr;62(4):1153-7. doi: 10.1002/art.27333. PMID 20131261
- [Background] Karnabi E, Qu Y, Wadgaonkar R, Mancarella S, Yue Y, Chahine M, Clancy RM, Buyon JP, Boutjdir M. Congenital heart block: identification of autoantibody binding site on the extracellular loop (domain I, S5-S6) of alpha(1D) L-type Ca channel. J Autoimmun. 2010 Mar;34(2):80-6. doi: 10.1016/j.jaut.2009.06.005. Epub 2009 Jul 28. PMID 19640679
- [Background] Reynolds HR, Buyon J, Kim M, Rivera TL, Izmirly P, Tunick P, Clancy RM. Association of plasma soluble E-selectin and adiponectin with carotid plaque in patients with systemic lupus erythematosus. Atherosclerosis. 2010 Jun;210(2):569-74. doi: 10.1016/j.atherosclerosis.2009.12.007. Epub 2009 Dec 16. PMID 20044088
- [Background] Saxena A, McDonnell E, Ramos PS, Sajuthi S, Marion MC, Langefeld CD, Buyon JP, Clancy RM. Preferential transmission of genetic risk variants of candidate loci at 6p21 from asymptomatic grandparents to mothers of children with neonatal lupus. Arthritis Rheum. 2012 Mar;64(3):931-9. doi: 10.1002/art.33366. PMID 22031281
- [Background] Izmirly PM, Saxena A, Kim MY, Wang D, Sahl SK, Llanos C, Friedman D, Buyon JP. Maternal and fetal factors associated with mortality and morbidity in a multi-racial/ethnic registry of anti-SSA/Ro-associated cardiac neonatal lupus. Circulation. 2011 Nov 1;124(18):1927-35. doi: 10.1161/CIRCULATIONAHA.111.033894. Epub 2011 Oct 3. PMID 21969015
- [Background] Briassouli P, Rifkin D, Clancy RM, Buyon JP. Binding of anti-SSA antibodies to apoptotic fetal cardiocytes stimulates urokinase plasminogen activator (uPA)/uPA receptor-dependent activation of TGF-beta and potentiates fibrosis. J Immunol. 2011 Nov 15;187(10):5392-401. doi: 10.4049/jimmunol.1101288. Epub 2011 Oct 17. PMID 22013113
- [Background] Routsias JG, Kyriakidis NC, Friedman DM, Llanos C, Clancy R, Moutsopoulos HM, Buyon J, Tzioufas AG. Association of the idiotype:antiidiotype antibody ratio with the efficacy of intravenous immunoglobulin treatment for the prevention of recurrent autoimmune-associated congenital heart block. Arthritis Rheum. 2011 Sep;63(9):2783-9. doi: 10.1002/art.30464. PMID 21618202
- [Background] Alvarez D, Briassouli P, Clancy RM, Zavadil J, Reed JH, Abellar RG, Halushka M, Fox-Talbot K, Barrat FJ, Buyon JP. A novel role of endothelin-1 in linking Toll-like receptor 7-mediated inflammation to fibrosis in congenital heart block. J Biol Chem. 2011 Sep 2;286(35):30444-30454. doi: 10.1074/jbc.M111.263657. Epub 2011 Jul 5. PMID 21730058
- [Background] Reed JH, Clancy RM, Purcell AW, Kim MY, Gordon TP, Buyon JP. beta2-glycoprotein I and protection from anti-SSA/Ro60-associated cardiac manifestations of neonatal lupus. J Immunol. 2011 Jul 1;187(1):520-6. doi: 10.4049/jimmunol.1100122. Epub 2011 May 20. PMID 21602492
- [Background] Reed JH, Clancy RM, Lee KH, Saxena A, Izmirly PM, Buyon JP. Umbilical cord blood levels of maternal antibodies reactive with p200 and full-length Ro 52 in the assessment of risk for cardiac manifestations of neonatal lupus. Arthritis Care Res (Hoboken). 2012 Sep;64(9):1373-81. doi: 10.1002/acr.21704. PMID 22511615
- [Background] Cherian TS, Kariuki SN, Franek BS, Buyon JP, Clancy RM, Niewold TB. Brief Report: IRF5 systemic lupus erythematosus risk haplotype is associated with asymptomatic serologic autoimmunity and progression to clinical autoimmunity in mothers of children with neonatal lupus. Arthritis Rheum. 2012 Oct;64(10):3383-7. doi: 10.1002/art.34571. PMID 22674082
- [Background] Izmirly PM, Buyon JP, Saxena A. Neonatal lupus: advances in understanding pathogenesis and identifying treatments of cardiac disease. Curr Opin Rheumatol. 2012 Sep;24(5):466-72. doi: 10.1097/BOR.0b013e328356226b. PMID 22832822
- [Background] Ramos PS, Marion MC, Langefeld CD; International Consortium on Systemic Lupus Erythematosus Genetics; Buyon JP, Clancy RM. Brief report: enrichment of associations in genes with fibrosis, apoptosis, and innate immunity functions with cardiac manifestations of neonatal lupus. Arthritis Rheum. 2012 Dec;64(12):4060-5. doi: 10.1002/art.34663. PMID 22886516
- [Background] Reed JH, Jain M, Lee K, Kandimalla ER, Faridi MH, Buyon JP, Gupta V, Clancy RM. Complement receptor 3 influences toll-like receptor 7/8-dependent inflammation: implications for autoimmune diseases characterized by antibody reactivity to ribonucleoproteins. J Biol Chem. 2013 Mar 29;288(13):9077-83. doi: 10.1074/jbc.M112.403303. Epub 2013 Feb 5. PMID 23386618
- See also: Research Registry for Neonatal Lupus Facebook Page — https://www.facebook.com/pages/Research-Registry-For-Neonatal-Lupus/212655652139338